CLINICAL TRIAL: NCT01150981
Title: Effect of Rosiglitazone on In-vivo Angiogenic Potential of Human Adipose Tissue
Brief Title: Effect of Rosiglitazone on the Vascular Biology of Human Fat Tissue
Acronym: RAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Samir Malkani, Study Principle Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12196
Record Dates: First submitted 2010-06-17; First posted 2010-06-25 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Metabolic Syndrome; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone (Experimental): One 8mg capsule daily for 6 weeks.
  Interventions: Drug: Rosiglitazone
- Placebo (Placebo Comparator): One capsule daily for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — One 8mg capsule daily for 6 weeks.
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Placebo — One capsule daily for 6 weeks.
  Arms: Placebo

SUMMARY:
Insulin resistance is a common condition that can lead to type 2 diabetes. One of the commonly prescribed diabetes medications, called rosiglitazone, works by decreasing insulin resistance. Rosiglitazone appears to work on fat cells. Animal studies suggest that rosiglitazone may work by increasing blood vessel growth in fat cells. The purpose of this research is to see if rosiglitazone also increases blood vessel growth in human fat cells. The investigators will compare results from before and after being on rosiglitazone for 6 weeks.

DETAILED DESCRIPTION:
Adipocytes play a crucial role in the control of metabolic homeostasis, by sequestering excess calories in the form of triglycerides, and secreting cytokines that control systemic fuel utilization. Sustained excess calorie consumption results in adipocyte hypertrophy and hyperplasia, and like any expanding tissue, requires increased capillary expansion to nourish the enlarged adipose tissue mass. Recent reports indicate that decreased capillary density in adipose tissue of obese individuals correlates with insulin resistance, suggesting that an imbalance of angiogenesis and adipogenesis may underlie this condition. To determine whether improvement in insulin sensitivity is related to changes in adipose tissue capillary development, we conducted a randomized, double-blind, placebo-controlled trial to determine capillary density, angiogenic growth potential, and metabolic parameters in healthy human volunteers before and after treatment with rosiglitazone, a potent insulin sensitizer.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight but otherwise in good general health.
2. Age 18 - 55 years.
3. Normal glucose tolerance.
4. Stable weight with BMI (27-44).
5. Stable medication use for the preceding month.
6. BP < 150/90.
7. Negative pregnancy test (*HCG), if female and of childbearing potential.
8. Practicing, and willing to continue to practice appropriate contraception throughout the study if a female of childbearing potential.

Exclusion Criteria:

1. Serious medical illness.
2. Pregnancy.
3. Tobacco use within the past 6 months.
4. Prior or current treatment with a thiazolidinedione.
5. Patients who have received an investigational drug in the past 30 days.
6. Use of systemic corticosteroids.
7. Known or suspected allergy to Rosiglitazone or any component of the preparation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Malkani, MD, Principal Investigator — UMass Worcester; Silvia Corvera, MD, Principal Investigator — UMass Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Gealekman O, Guseva N, Gurav K, Gusev A, Hartigan C, Thompson M, Malkani S, Corvera S. Effect of rosiglitazone on capillary density and angiogenesis in adipose tissue of normoglycaemic humans in a randomised controlled trial. Diabetologia. 2012 Oct;55(10):2794-2799. doi: 10.1007/s00125-012-2658-2. Epub 2012 Jul 31. PMID 22847059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates of recruitment January 2007 to January 2010
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 20 | 15
Completed | 16 | 13
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 20 | 15 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 35
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.25 (2.42) | 40.2 (10.23) | 40.09 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Adipose Tissue Capillary Sprout Formation
Description: Adipose tissue collected at 8 weeks was cut into ~1mm pieces which were embedded in individual wells of a 96 well plate containing growth factor depleted Matrigel. Wells were filled with media supplemented with endothelial growth factors, replaced every second day. Values for each patient are expressed as the difference in the average number of capillary branches (sprouts) formed by each of approximately 50 explants between day 14 and day 7. The number of branches forming on the periphery (defined as at least three cells in a branch structure) was counted by two investigators at day 7 and 14.
Time Frame: 8 weeks
Population: The number of subjects was based on the power of calculations in being able to demonstrate a difference from baseline in fat tissue microvasculature, change in HOMA2 and serum adiponectin after 6 weeks of rosiglitazone intake in all groups.
Measure: Mean (Standard Deviation); unit: number of capillary sprouts
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 16 | 13
number of capillary sprouts | 143.5 (41.12) | 122.1 (43.88)

2. Secondary Outcome: Serum Adiponectin
Description: Adiponectin concentrations in serum were measured in ng/ml, in both arms at baseline and at 8 weeks, i.e. 2 weeks after stopping drug or placebo treatment
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 16 | 13
ng/ml | 28.56 (2.89) | 14.64 (2.86)

ADVERSE EVENTS:
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No